CLINICAL TRIAL: NCT03272360
Title: A Prospective Sample Collection Study in Patients With Pelvic Pain Undergoing Laparoscopy for Biomarker Identification in Endometriosis
Brief Title: Endometriosis Biomarker Discovery Study
Acronym: EMBARK
Status: Withdrawn | Type: Observational
Why Stopped: company decision to suspend project
Sponsor: Myriad Genetic Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EP-002
Record Dates: First submitted 2016-09-06; First posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2016-09

CONDITIONS: Chronic Pelvic Pain; Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma, whole blood, urine, and endometrial tissue

GROUPS / COHORTS (2):
- Chronic Pelvic Pain
- Elective Tubal Ligation

SUMMARY:
This is a prospective, Single time point, discovery study intending to identify biomarkers that can differentiate endometriosis from other underlying reasons for pelvic pain. Patients undergoing laparoscopy for evaluation of chronic pelvic pain or elective tubal ligation will be enrolled for collection of tissue samples at the time of laparoscopy.

DETAILED DESCRIPTION:
This study will be a prospective collection of blood, urine, and endometrial tissue from women with chronic pelvic pain symptoms, with or without infertility, who require evaluation by laparoscopy. Women undergoing laparoscopy for elective tubal ligation will also be investigated similarly and serve as the negative control. Subjects will be queried regarding sociodemographic characteristics, medical and reproductive history, pain and lifestyle as well as assessment for differential diagnoses such as interstitial cystitis and idiopathic bowel syndrome. Endometriosis severity will be captured by rASRM staging during laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give informed consent.
2. Aged 18-45 years old who has a regular menstrual cycle (26 to 32 days in length).
3. Undergoing a planned diagnostic or therapeutic laparoscopy for the indication of pelvic pain or for elective tubal ligation.
4. One prior pregnancy for tubal ligation patients.

Exclusion Criteria:

1. Prior surgical diagnosis of endometriosis.
2. Currently pregnant or breastfeeding.
3. Clinical suspicion of pelvic inflammatory disease (PID) or urinary tract infection.
4. Current malignancy except non-melanoma skin cancer adequately treated.
5. Known major systemic disease, including but not limited to inflammatory disease, autoimmune disease.
6. Use of immunosuppressants in the past 3 months.
7. Use of injectable reproductive hormonal therapy within the past 3 months and have not menstruated since last dose.
8. If reproductive hormonal implant has been used in the past, it must have been removed > 3 months prior to study entry and subject must have menstruated since removal.
9. Use of intrauterine device (IUD) in the past 3 months.
10. Use of any other reproductive hormone therapy within the past 3 months, except for oral contraceptives (OCPs).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women seeking care at OB/GYN clinics and fertility centers
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
The identification of biomarker(s) that are differentially expressed in endometriosis in the context of pelvic pain | Baseline (pre-operative)
  The primary variables will be the DiscoveryMAP analytes identified in blood and/or urine and the mRNA transcriptome in endometrial tissue. DiscoveryMAP is a comprehensive, quantitative platform of immunoassays evaluating multiple analytes in various body system categories: cytokines, chemokines, metabolic markers, hormones, growth factors, tissue remodeling proteins, angiogenesis markers, acute phase reactants, and cancer markers

SECONDARY OUTCOMES:
The identification of biomarker(s) that are associated with endometriosis severity | Baseline (pre-operative)
  The secondary variables will be measures of endometriosis severity: rASRM staging of endometriosis and pain severity from clinical survey